CLINICAL TRIAL: NCT01481415
Title: Left Atrial Volume and Function in Healthy Children Assessed by Three Dimensional Echocardiography
Brief Title: Left Atrial Volume and Function in Children Assessed by Echo 3DRT: Reference Values for Normal Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Laise Antonia Bonfim Guimaraes, Dr, Hospital Israelita Albert Einstein
Other Study IDs: p1
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Left Ventricular Function Good
Keywords: left atrial; three-dimensional echocardioraphy; left atrial function

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators study is trying to find the normal value to left atrial volume and left atrial function in healthy children by tridimensional real time echocardiography avaluation.

ELIGIBILITY:
Inclusion Criteria:

* research murmur

Exclusion Criteria:

* any congenital heart disease
* any systemic disease

Ages: 3 Months to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2011-11; Primary Completion 2011-11 (Actual); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Laise Antonia Bonfim Guimaraes, MD, Principal Investigator — Sociedade Beneficente Israelita Albert Einstein
Locations (2):
- Brazil (2):
  - Hospital Israelita Albert Einstein, Sâo Paulo, Sao Pauo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo